CLINICAL TRIAL: NCT04459806
Title: Evaluation of Intracranial Pressure Time Dose by the New Integra CereLink ICP Monitor
Brief Title: Intracranial PrEssure Time dOse (ImPETO)
Acronym: ImPETO
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: ImPETO
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Intracranial Hypertension; Traumatic Brain Injury; Subarachnoid Hemorrhage; Intracranial Hemorrhages
MeSH Terms: conditions — Intracranial Hypertension; Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Intracranial Hemorrhages

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: intracranial pressure monitoring — Invasive monitoring of intracranial pressure by using CereLink monitor.

SUMMARY:
The new Integra CereLink ICP monitor integrate the possibility of recording and displaying continuously the AUC (Pressure Time Dose, PTD) and other ICP derived variables and provide the possibility of evaluating the utility of this information at the bedside. It offers the opportunity to test in a standardized way the clinical value of the PTD computation in this setting.

Therefore, this study aims to test clinically if PTD recorded continuously is associated to patients' outcome and to identify a threshold of PTD associated with the transition from good to negative outcomes.

DETAILED DESCRIPTION:
Intracranial pressure (ICP) monitoring is the most common neuromonitoring modality used in neurocritical care (NCCU). Its application both as a stand-alone monitoring or in association with other systems (brain oxygenation, brain microdialysis, electroencephalography, transcranial Doppler ultrasound, etc.) has several indications, which rely on local, national policies, and international guidelines. In 2014, ESICM with the Neurocritical Care Society released a multidisciplinary Consensus Statement to provide a guidance on Multimodality Monitoring in Neurocritical Care, including ICP: "ICP and CPP monitoring are recommended as a part of protocol-driven care in patients who are at risk of elevated intracranial pressure based on clinical and/or imaging features. (Strong recommendation, moderate quality of evidence)". The most recent Brain Trauma Foundation guidelines focused on the importance of ICP monitoring, especially in severe traumatic brain injury, but a living systematic review showed that the compliance rate to these guidelines was low (31%; range 18-83%). Most of the ICP monitoring guidance orbits around traumatic brain injury, while there are uncertainties around indication of ICP monitoring in non-traumatic brain injury (acute subarachnoid hemorrhage and intracerebral hemorrhage).

Similarly, ICP thresholds, threshold-based treatment strategies and their impact on outcome have not been established yet. The interpretation of data on ICP practice has a limited value without some reference to the intensity of therapy directed at control of ICP. The Therapy Intensity Level (TIL) may be a more sensitive measure of the severity of pathophysiology but the effect on outcome of existing differences in practice is unclear.

In most intensive care units, ICP values are summarized hourly in bedside charts by trained nurses, as end-hour ICP, and similar data have been used in large randomized clinical trials testing neuroprotective treatments for TBI patients.

However, several single center studies showed that this manual acquisition method is suboptimal and could miss episodes of high ICP compared to high-resolution, computerized acquisition systems. Computers allow also the computation offline of ICP derived parameters. Vik proposed that the degree of ICP above the treatment threshold can be estimated by the area under the curve (AUC) of ICP versus time in patients with TBI, i.e. the "ICP dose". A significant relationship between the ICP dose, the worst Marshall CT score, and patient outcome exists, suggesting that the AUC method may be useful in refining and improving the treatment of ICP in patients with TBI. Moreover, small cohort studies confirmed this relationship between the dose of ICP and patient outcome, suggesting that the dose of ICP may be useful in refining and improving the treatment of ICP in patients with TBI. In a single centre cohort TBI study, increased ICP dose was associated with mortality and poor functional outcome at 6 months. However, there was no association between episodic ICP data and outcome, proposing this index as candidate "biomarker" of the disease.

Even if the concept is attracting, all these computations have been collected a posteriori and no single ICP monitoring system was able to display the ICP dose continuously, making it useful at the bedside.

The new Integra CereLink ICP monitor integrate the possibility of recording and displaying continuously the AUC (Pressure Time Dose, PTD) and other ICP derived variables and provide the possibility of evaluating the utility of this information at the bedside. It offers the opportunity to test in a standardized way the clinical value of the PTD computation in this setting.

Therefore, the study aims to test clinically if PTD recorded continuously is associated to patients' outcome and to identify a threshold of PTD associated with the transition from good to negative outcomes.

Hypothesis:

* High PTD is associated with worse outcome.
* A threshold of PTD associated with good outcomes (mortality and 6 months outcome) might be identified.
* A better PTD summary report, more closely associated with outcome, will make this parameter useful at the bedside.

Methods:

The study is prospective, observational, international cohort study in centers already using the new Integra CereLink ICP monitor (released in spring 2019).

Treatments and clinical decisions will not be affected by the participation to the protocol that is purely observational.

Potential centers involved are listed in the Addendum.

Each investigator will notify the relevant ethics committee, in compliance with the local legislation and rules. Since patients recruited in this study will not be able to provide an informed consent at the time of recruitment (patient in coma requiring ICP monitoring), the responsible clinical/research staff will act as Consultee and consent eligible patients after discussion with the next-of-kin. At follow-up, patients who have regained capacity will be asked to provide Informed Consent for the acute data and follow-up or deny research participation and request destruction of acute data collected.

Data collection will be web-based. Participating centres will register electronically and collect data via an electronic Case-Report Form (RedCAP) and data will be anonymized locally. The data resides at the University Milano-Bicocca; all procedures will comply with the EU regulation on data protection 2016/679 on the protection of natural persons regarding personal data processing and movement.

A reduced set of demographic characteristics, past medical history information, diagnosis, timeline, clinical presentation of ABI and administered treatments will be extracted from patients' medical records.

ICP high-resolution data will be downloaded from the Integra CereLink ICP monitor:

1. mean ICP;
2. ICP dose. Centres will collect mortality and GOSE at ICU/hospital discharge and GOSE at 6 months. The GOSE at the End-of-Study will be collected via phone structured interviews to patients and/or family members using a validated questionnaire.

Data accuracy will be verified automatically in the database through validity and consistency checks on relevant variables and, additionally, a trained staff at the University of Milano-Bicocca in Monza will periodically perform checks of completeness and consistency of the information to ensure data quality.

Statistical plan:

Descriptive statistics will be used to summarize demographic, clinical features and outcomes. Kaplan-Maier estimates will be used to describe mortality and the Cox model to assess the association with PTD adjusting for potential confounders. The shared frailty joint model will be used to assess the predictiveness of the longitudinal PTD profile on mortality. The logistic model will be used to assess the role of PTD on GOSE dichotomized as poor and good outcome (poor outcome GOSE: 1-4; good outcome GOSE: 5-8). All tests will be two-sided with a significant level of 0.05.

No formal sample size calculation was performed but based on the potentiality of recruitment of the centers involved in the study, we expect to enrol at least 200 patients (with an average of 15 patients per center).

Expected results:

* The PTD (Pressure Time Dose) recorded by the Integra CereLink ICP monitor is related with outcome. Higher PTD are associated with worse outcomes.
* The max PTD associated with good outcomes will be estimated.
* The Investigators aim to identify the best way of summarizing PDT for clinical use.
* To demonstrate that PTD is a better predictor of outcome compared with end-hour ICP values (standard now)

Ethical aspects:

This is a prospective observational cohort study: no additional costs will be attribute to the Insitution/s.

Data collection will be web-based. Participating centres will collect data via an electronic Case-Report Form (REDCAP cloud); data will be automatically pseudoanonymized with a numeric alpha code; the list of correspondence between the patient's code and its identity will be stored in a safe place and access to this data will be granted only to study PI and study staff delegated by the PI and listed in the delegation log. The data resides at the University of Milano-Bicocca. The study will be conducted in accordance with the Helsinki Declaration and in accordance with the rules of Good Clinical Practice (D.M. Healthcare of 15/07/1997 and s.m.i.) as well as with the applicable regulatory provisions.

The patient's personal data will be processed in accordance with the European Personal Data Protection Regulation (GDPR), Di.Lgs. 196/2003 and subsequent changes and additions, and any other Italian law applicable to the protection of personal data (from which it later defined as "applicable data protection law").

The roles and responsibilities related to the project will be explained in a further and separate act between the Promoter and the institution.

There are no physical, psychical or social risks for the patients enrolled as the study is based on a prospective analysis of clinical data. Being that, in Italy, no informed consent forms will be submitted to patient according to AIFA Guidelines (Determinazione del 20 Marzo 2008, G.U. n.76 del 31/03/2008 - Linee guida per la classificazione e conduzione sugli studi osservaziona/i sui farmaci) but only a privacy statement will be submitted to patients that the local investigator will be able to re-contact. Being a retrospective analysis, all the IRB related procedures will be managed following the local laws.

The study will be conducted according to Helsinki Declaration and to Good Clinical Practice (D.M. Sanità del 18/07/1997 e s.m.i.).

Data property:

The Promoter has the property of the study database, study execution and results. Study results will be published by autonomous decision by the Promoter. The Promoter is committed to publish the results of the study.

Publication on a peer reviewed journal:

The Investigators aim a publication on a peer reviewed journal. A writing committee, composed in part of the SC members, will draft the work and the SC members will be authors of the manuscript. Additional authorship of the main manuscript will follow the International Committee of Medical Journal Editors (ICMJE) recommendations. For each centre, a participant will be indicated in the group authorship list.

Funding:

A financial support will be made available by Integra Lifesciences project (43.000€) for statistical analyses, data management and eCRF development.

ELIGIBILITY:
Inclusion Criteria:

* Aged within 18 and 80 years;
* Diagnosed of an acute brain injury (ABI) for hemorrhagic stroke (including intracerebral hematoma or subarachnoid hemorrhage) or traumatic brain injury;
* ICP monitoring started for clinical indication and accordingly to local policies
* ICP device connected to the Integra CereLink ICP monitor.

Exclusion Criteria:

* ICP monitoring not inserted
* No availability of the Integra CereLink ICP monitor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute brain injury (ABI) due to hemorrhagic stroke (including intracerebral hematoma or subarachnoid hemorrhage) or traumatic brain injury.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between PTD and in-hospital mortality. | 12 months
  To assess the association between PTD and in-hospital mortality.

SECONDARY OUTCOMES:
Association between PTD and 6 months GOSE | 12 months
  To assess the association between PTD and 6 months GOSE (Glasgow Outcome Scale extended).
PTD summary measure. | 12 months
  To identify the PTD summary measure (e.g. mmHg/h max, mmHg/day, mmHg/week) that maximize the outcome prediction.
Outcome predictiveness of PTD and end hour ICP. | 12 months
  To compare the outcome predictiveness of PTD and end hour ICP.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, Professor, Principal Investigator — University of Milano Bicocca
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, MB, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Roux P, Menon DK, Citerio G, Vespa P, Bader MK, Brophy GM, Diringer MN, Stocchetti N, Videtta W, Armonda R, Badjatia N, Boesel J, Chesnut R, Chou S, Claassen J, Czosnyka M, De Georgia M, Figaji A, Fugate J, Helbok R, Horowitz D, Hutchinson P, Kumar M, McNett M, Miller C, Naidech A, Oddo M, Olson D, O'Phelan K, Provencio JJ, Puppo C, Riker R, Robertson C, Schmidt M, Taccone F. Consensus summary statement of the International Multidisciplinary Consensus Conference on Multimodality Monitoring in Neurocritical Care: a statement for healthcare professionals from the Neurocritical Care Society and the European Society of Intensive Care Medicine. Neurocrit Care. 2014 Dec;21 Suppl 2(Suppl 2):S1-26. doi: 10.1007/s12028-014-0041-5. PMID 25208678
- [Background] Carney N, Totten AM, O'Reilly C, Ullman JS, Hawryluk GW, Bell MJ, Bratton SL, Chesnut R, Harris OA, Kissoon N, Rubiano AM, Shutter L, Tasker RC, Vavilala MS, Wilberger J, Wright DW, Ghajar J. Guidelines for the Management of Severe Traumatic Brain Injury, Fourth Edition. Neurosurgery. 2017 Jan 1;80(1):6-15. doi: 10.1227/NEU.0000000000001432. PMID 27654000
- [Background] Cnossen MC, Scholten AC, Lingsma HF, Synnot A, Tavender E, Gantner D, Lecky F, Steyerberg EW, Polinder S. Adherence to Guidelines in Adult Patients with Traumatic Brain Injury: A Living Systematic Review. J Neurotrauma. 2021 Apr 15;38(8):1072-1085. doi: 10.1089/neu.2015.4121. Epub 2016 Aug 25. PMID 26431625
- [Background] Helbok R, Olson DM, Le Roux PD, Vespa P; Participants in the International Multidisciplinary Consensus Conference on Multimodality Monitoring. Intracranial pressure and cerebral perfusion pressure monitoring in non-TBI patients: special considerations. Neurocrit Care. 2014 Dec;21 Suppl 2:S85-94. doi: 10.1007/s12028-014-0040-6. PMID 25208677
- [Background] Chesnut RM, Bleck TP, Citerio G, Classen J, Cooper DJ, Coplin WM, Diringer MN, Grande PO, Hemphill JC 3rd, Hutchinson PJ, Le Roux P, Mayer SA, Menon DK, Myburgh JA, Okonkwo DO, Robertson CS, Sahuquillo J, Stocchetti N, Sung G, Temkin N, Vespa PM, Videtta W, Yonas H. A Consensus-Based Interpretation of the Benchmark Evidence from South American Trials: Treatment of Intracranial Pressure Trial. J Neurotrauma. 2015 Nov 15;32(22):1722-4. doi: 10.1089/neu.2015.3976. Epub 2015 Aug 31. PMID 26061135
- [Background] Hemphill JC 3rd, Greenberg SM, Anderson CS, Becker K, Bendok BR, Cushman M, Fung GL, Goldstein JN, Macdonald RL, Mitchell PH, Scott PA, Selim MH, Woo D; American Heart Association Stroke Council; Council on Cardiovascular and Stroke Nursing; Council on Clinical Cardiology. Guidelines for the Management of Spontaneous Intracerebral Hemorrhage: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2015 Jul;46(7):2032-60. doi: 10.1161/STR.0000000000000069. Epub 2015 May 28. PMID 26022637
- [Background] Chesnut R, Videtta W, Vespa P, Le Roux P; Participants in the International Multidisciplinary Consensus Conference on Multimodality Monitoring. Intracranial pressure monitoring: fundamental considerations and rationale for monitoring. Neurocrit Care. 2014 Dec;21 Suppl 2:S64-84. doi: 10.1007/s12028-014-0048-y. PMID 25208680
- [Background] Guiza F, Depreitere B, Piper I, Citerio G, Chambers I, Jones PA, Lo TY, Enblad P, Nillson P, Feyen B, Jorens P, Maas A, Schuhmann MU, Donald R, Moss L, Van den Berghe G, Meyfroidt G. Visualizing the pressure and time burden of intracranial hypertension in adult and paediatric traumatic brain injury. Intensive Care Med. 2015 Jun;41(6):1067-76. doi: 10.1007/s00134-015-3806-1. Epub 2015 Apr 18. PMID 25894624
- [Background] Vik A, Nag T, Fredriksli OA, Skandsen T, Moen KG, Schirmer-Mikalsen K, Manley GT. Relationship of "dose" of intracranial hypertension to outcome in severe traumatic brain injury. J Neurosurg. 2008 Oct;109(4):678-84. doi: 10.3171/JNS/2008/109/10/0678. PMID 18826355
- [Background] Magni F, Pozzi M, Rota M, Vargiolu A, Citerio G. High-Resolution Intracranial Pressure Burden and Outcome in Subarachnoid Hemorrhage. Stroke. 2015 Sep;46(9):2464-9. doi: 10.1161/STROKEAHA.115.010219. Epub 2015 Aug 4. PMID 26243224
- [Background] Stocchetti N, Maas AI. Traumatic intracranial hypertension. N Engl J Med. 2014 Sep 4;371(10):972. doi: 10.1056/NEJMc1407775. No abstract available. PMID 25184881
- [Background] Shutter LA, Timmons SD. Intracranial Pressure Rescued by Decompressive Surgery after Traumatic Brain Injury. N Engl J Med. 2016 Sep 22;375(12):1183-4. doi: 10.1056/NEJMe1609722. Epub 2016 Sep 7. No abstract available. PMID 27604048
- [Background] Yuan Q, Wu X, Sun Y, Yu J, Li Z, Du Z, Mao Y, Zhou L, Hu J. Impact of intracranial pressure monitoring on mortality in patients with traumatic brain injury: a systematic review and meta-analysis. J Neurosurg. 2015 Mar;122(3):574-87. doi: 10.3171/2014.10.JNS1460. Epub 2014 Dec 5. PMID 25479125
- [Background] Stocchetti N, Carbonara M, Citerio G, Ercole A, Skrifvars MB, Smielewski P, Zoerle T, Menon DK. Severe traumatic brain injury: targeted management in the intensive care unit. Lancet Neurol. 2017 Jun;16(6):452-464. doi: 10.1016/S1474-4422(17)30118-7. PMID 28504109
- [Background] Zanier ER, Ortolano F, Ghisoni L, Colombo A, Losappio S, Stocchetti N. Intracranial pressure monitoring in intensive care: clinical advantages of a computerized system over manual recording. Crit Care. 2007;11(1):R7. doi: 10.1186/cc5155. PMID 17233895
- [Background] Sheth KN, Stein DM, Aarabi B, Hu P, Kufera JA, Scalea TM, Hanley DF. Intracranial pressure dose and outcome in traumatic brain injury. Neurocrit Care. 2013 Feb;18(1):26-32. doi: 10.1007/s12028-012-9780-3. PMID 23055087